CLINICAL TRIAL: NCT00171782
Title: Valsartan Plus Hydrochlorothiazide in Patients With Hypertension and Cardiovascular Risk Factors
Brief Title: Hypertension and Cardiovascular Risk Factors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAH631BCO02
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: HYPERTENSION
Keywords: HYPERTENSION; VALSARTAN; VALSARTAN AND HYDROCHLOROTHIAZIDE; RISK FACTORS
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Drug: VALSARTAN+HYDROCHLOROTHIAZIDE

SUMMARY:
A study to evaluate the efficacy of valsartan+chydochlorothiazide in patients with stage 2 hypertension and cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* - Patients who give consent
* Men and women 18 to 80 years of age
* Patients with hypertension (systolic >159 mm, diastolic >100 mm)
* Patients meeting laboratory criteria

Exclusion Criteria:

* - Pregnant women
* Women not using approved contraception methods
* Secondary hypertension

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2004-02; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline systolic blood pressure at 8 weeks

SECONDARY OUTCOMES:
Blood pressure less than 140/90 mmHg at 8 weeks
Reduction from baseline in diastolic blood pressure greater than or equal to 10 mmHg
Reduction from baseline in systolic blood pressure greater than or equal to 20 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals